CLINICAL TRIAL: NCT04360941
Title: PAveMenT: Phase Ib Study of Palbociclib and Avelumab in Metastatic AR+ Triple Negative Breast Cancer
Brief Title: PAveMenT: Palbociclib and Avelumab in Metastatic AR+ Triple Negative Breast Cancer
Acronym: PAveMenT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Pfizer (Industry); Breast Cancer Now (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCR4884
Record Dates: First submitted 2020-04-07; First posted 2020-04-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer; Locally Advanced Breast Cancer; Recurrent Breast Cancer; Metastatic Breast Cancer; ER+ Breast Cancer; HER2-positive Breast Cancer
Keywords: Palbociclib; Avelumab; Measurable Disease; Inoperable Disease
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — palbociclib; avelumab

STUDY DESIGN:
Intervention Model Description: This is a two-part phase 1b trial of induction palbociclib with the addition of avelumab. In Part A of the study, the MTD of the study will be determined using a 3+3 design. There will be a 1-week interval between the first and second patients started at each dose level.
  In Part B, the MTD dose level will be expanded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Two-part phase 1b trial of induction palbociclib with avelumab (Experimental): Recruitment to Part A will be conducted at the Royal Marsden Hospital only. Up to 18 patients will be recruited for dose escalation of palbociclib in combination with fixed dose avelumab.
  Part B will recruit at up to 8 high volume centres. Up to 27 patients will be recruited to treatment with the maximum tolerated dose and schedule established in part A. In Part B of the study, additional selection by triple negative histology and positive androgen receptor status will define the study population.
  Interventions: Drug: Palbociclib; Drug: Avelumab

INTERVENTIONS:
Drug: Palbociclib — Highly selective oral inhibitor of CDK4 and CDK6.
  Other Names: Ibrance
Drug: Avelumab — Fully human IgG1 monoclonal antibody (mAb) binds to the PD-L1 cell surface ligand and blocks its interaction with the PD-1 cell surface receptor.
  Other Names: Bavencio

SUMMARY:
This clinical study is aiming to determine the safest doses and schedule for the combination of two drugs named palbociclib and avelumab.

The study will also be investigating how effective the combination is for a subgroup of breast cancer patients whose cancer expresses the androgen receptor (AR) but not the oestrogen (hormone) or HER2 receptors. Palbociclib is a drug used in routine care for hormone-receptor (HR) positive and HER2 negative advanced breast cancer, the most common subtype of breast cancer.

It is possible that the combination of palbociclib and avelumab will be a more effective cancer treatment than each drug separately, but this is unknown and this study is needed to establish the best dosage and schedule of each drug as well as how effective the combination is.

DETAILED DESCRIPTION:
This is a phase Ib study designed to confirm the safety and evaluate the efficacy of palbociclib combined with avelumab in AR positive TNBC. It is a multi-centre study design (it will run at several hospitals in the UK).

Palbociclib inhibits two proteins involved in cell growth called cyclin dependent kinase 4 and cyclin dependent kinase 6 (CDK4/6). Inhibiting CDK4/6 stops cells, such as cancer cells, from dividing and multiplying further. Palbociclib is currently approved for the treatment of metastatic HR positive HER2 negative breast cancer, based on good results from large clinical trials. Laboratory studies have shown that palbociclib might be also useful in some patients with triple negative breast cancer, an aggressive subtype of breast cancer that does not express the hormone receptors or HER2 receptor, but only if the cancer is positive for the androgen-receptor (AR).

Avelumab is an immunotherapy drug which does not destroy cancer cells, but tries to stimulate the body's immune system to do this. Avelumab has been tested in a number of different types of tumours including breast cancer, but although approved for use in the USA, it is not currently an approved standard treatment in the UK. The combination of both drugs has never been tested in humans before.

Recruitment to Part A will be conducted only at the Royal Marsden Hospital and Part A of the study will establish the maximum tolerated dose (MTD) and optimal schedule of the combination in any suitable patients with advanced breast cancer. Once this dose schedule has been confirmed, the chosen dose level will be recruited to, aiming to include 27 patients with AR positive TNBC (Part B).Part B will recruit at up to 8 high volume centres. The androgen receptor is not routinely tested for in hospital laboratories, so patients with advanced triple negative breast cancer who are interested in taking part in the study will be asked to provide consent for previously taken cancer samples/biopsies to be sent to the Royal Marsden for testing, to see if the cancer expresses the androgen receptor, which would make participants potentially eligible for part B of the study. Approximately 20% of triple negative breast cancers express AR. This phase of the study will include important translational work using new cancer samples (biopsies) and blood samples to investigate potential "biomarkers" -predictors of efficacy and resistance to the combination.

In Part A of the study, patients with previously treated, advanced breast cancer will have an ECG (heart trace) a CT scan of the body and potentially an MRI scan of the brain and a bone scan (depending upon where the breast cancer is known to have spread to) as well as blood tests to determine if participants are suitable for the study.

During the study participants will receive daily palbociclib tablets and intravenous infusions of avelumab every two weeks. Participants will be monitored with regular blood tests and repeat CT scans every 8 weeks. At whatever time point the treatment stops working, the patient will stop treatment and will be asked to have further blood tests one month later as well as a check up with the study doctor.

In Part B of the study, patients with triple negative histology and positive androgen receptor status tested at the Royal Marsden will be required to have a cancer biopsy before participants start treatment on the study. LIke in Part A, participants will also have an ECG (heart trace)a CT scan of the body and potentially an MRI scan of the brain and a bone scan (depending upon where the breast cancer is known to have spread to) as well as blood tests to determine if participants are suitable for the study. During the study participants will receive daily palbociclib tablets and intravenous infusions of avelumab every two weeks. Participants will be monitored with regular blood tests and check-ups with the study doctor and repeat CT scans every 8 weeks as well as additional blood tests for research. After 3 weeks of treatment, the patient may have a further tumour biopsy, which is optional. At whatever timepoint the treatment stops working, the patient will stop treatment and will be asked to have further blood tests and a further biopsy. Participants will also have a check-up with the study doctor and blood tests one month later.

A maximum of 45 breast cancer patients will be enrolled; up to 18 patients in part A and 27 patients with AR+ triple negative breast cancer in part B.

ELIGIBILITY:
Inclusion Criteria Part A:

1. Patients with recurrent inoperable locally advanced or metastatic breast cancer.
2. Previously treated with at least one prior line of chemotherapy for advanced disease, but no more than two prior lines of chemotherapy for advanced disease. Patients with ER+ breast cancer must have received at least one prior line of hormone therapy for advanced disease. Patients with HER2+ breast cancer must have received at least one prior line of HER2 directed therapy.
3. Measurable disease (RECIST 1.1)
4. Haematological and biochemical indices within the ranges stated in the study protocol. These measurements must be performed within one week (Day -7 to Day 1) before the patient goes in the trial.
5. Women/female patients with child-bearing potential (defined as the fertile status following menarche and until becoming post-menopausal unless permanently sterile by methods that include hysterectomy, bilateral salpingectomy and bilateral oophorectomy) must have a negative urine or serum pregnancy test within 7 days prior to start of trial.

   Women/females of child bearing potential or their male partners must use a highly effective method of contraception for 2 weeks before starting the study treatment, throughout the treatment period and for 1 month after discontinuation of treatment with palbociclib and avelumab (women/female patients) or 14 weeks (men/male patients). Highly effective methods are defined as methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods, such methods include:
   * Oral, intra-vaginal or transdermal combined hormonal contraception
   * Oral, injectable or implantable progesterone-only contraception
   * Intrauterine device
   * Intrauterine hormone-releasing system,
   * Bilateral tubal occlusion
   * Vasectomised partner
   * True abstinence:* When this is in line with the preferred and usual lifestyle of the subject

   Key: * it is only considered highly effective if the patient is refraining from sexual intercourse during the entire period of risk associated with the study treatments
6. 18 years of age or over.
7. World Health Organisation (WHO) performance status 0 or 1
8. Estimated life expectancy of at least 3 months in the opinion of the investigator
9. Signed and dated informed consent.
10. Patients willing and able to comply with scheduled visits, treatment plans, laboratory tests, follow up and other procedures

Inclusion Criteria Part B:

1. Patients with recurrent inoperable locally advanced or metastatic AR+ triple negative breast cancer with ER, PgR and HER2 status determined locally and AR determined centrally on archival metastatic tissue. Archival tissue from the primary tumour (which must have been ER/PgR negative and collected within 5 years prior to metastatic relapse) may be used for AR testing if no archival metastatic tissue is available.
2. Previously treated with at least one prior line of chemotherapy for advanced disease, but no more than two prior lines of chemotherapy for advanced disease.
3. Measurable disease (RECIST 1.1) amenable to fresh biopsy
4. Haematological and biochemical indices within the ranges stated in the study protocol. These measurements must be performed within one week (Day -7 to Day 1) before the patient goes in the trial.
5. Female patients with child-bearing potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.

   Women/females of child bearing potential or their male partners must use a highly effective method of contraception for 2 weeks before starting the study treatment, throughout the treatment period and for 1 month after discontinuation of treatment with palbociclib and avelumab (women/female patients) or 14 weeks (men/male patients). Highly effective methods are defined as methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods, such methods include:
   * Oral, intra-vaginal or transdermal combined hormonal contraception
   * Oral, injectable or implantable progesterone-only contraception
   * Intrauterine device
   * Intrauterine hormone-releasing system,
   * Bilateral tubal occlusion
   * Vasectomised partner
   * True abstinence:* When this is in line with the preferred and usual lifestyle of the subject

   Key: * it is only considered highly effective if the patient is refraining from sexual intercourse during the entire period of risk associated with the study treatments
6. Age 18 years of age or over
7. World Health Organisation (WHO) performance status 0 or 1
8. Estimated life expectancy of at least 3 months in the opinion of the investigator
9. Signed and dated informed consent
10. Patients willing and able to comply with scheduled visits, treatment plans, laboratory tests, follow up, and other procedures
11. Available archival breast primary tumour tissue (or metastatic tissue if de novo metastatic disease)
12. Patient willing to undergo a mandatory baseline fresh tumour tissue biopsy procedure (clinical or radiologically-guided)

Exclusion Criteria Parts A & B:

1. Oral chemotherapy within two weeks, weekly iv chemotherapy within three weeks or any other systemic chemotherapy or investigational medicinal products during the previous four weeks.
2. Hormonal therapy within 7 days except luteinizing hormone-releasing hormone (LHRH) analogues for ovarian suppression. Bisphosphonates or RANK ligand antagonists are permitted for the management of bone metastases.
3. Previous exposure to immune checkpoint inhibitors or immune co-stimulatory drugs in the advanced setting. (Note: Patients who have received neoadjuvant and/or adjuvant pembrolizumab are eligible if treatment was completed at 6 months prior to metastatic relapse.)
4. Previous treatment with palbociclib or any agents which inhibit CDK4/6. (Note: Patients who have received adjuvant abemaciclib or ribociclib for early breast cancer are eligible if treatment was completed at least 12 months prior to metastatic relapse.)
5. Major surgery (excluding minor procedures, e.g. placement of vascular access) within 4 weeks or radiation therapy within 14 days prior to study entry
6. Patients with known symptomatic brain metastases requiring steroids, untreated brain metastases, leptomeningeal disease or spinal cord compression.
7. Active infection requiring systemic therapy
8. Any of the following within 12 months prior to study entry: myocardial infarction, history of myocarditis, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack.
9. Uncontrolled hypertension or cardiac dysrhythmia including atrial fibrillation
10. Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
11. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
12. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis (even if fully resolved), pulmonary fibrosis, end stage renal disease on haemodialysis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
13. Patients on warfarin or direct acting oral anticoagulants. Patients requiring anticoagulation for rate-controlled AF or previous venous thromboembolism should be switched to low-molecular weight heparin.
14. Known HIV or AIDS-related illness, active infection requiring systemic therapy, or positive HBV or HCV test indicating acute or chronic infection
15. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI CTCAE v 5), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
16. Inability or unwillingness to swallow pills, or receive IV injections.
17. Persisting toxicity related to prior therapy >Grade 1 (except for stable peripheral neuropathy grade ≤2 or alopecia grade ≤2).
18. Pregnancy or lactation (women/females of childbearing potential must have a negative pregnancy test within 7 days prior to treatment initiation)
19. Diagnosis of other malignancy within 3 years, except for previous breast cancer, adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix, or low-grade (Gleason ≤6) prostate cancer
20. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this study. Participation in an observational trial would be acceptable.
21. Known prior or suspected hypersensitivity to investigational products or to any of the excipients
22. Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines. Live vaccines must also be avoided for 3 months after the last dose of avelumab.
23. Any psychiatric condition that would prohibit the understanding or rendering of informed consent
24. Requirement for continued use of preparations containing St. John's Wort is specifically contraindicated. Other herbal medicinal or natural products that patient is intended to take during the trial must be explored at the beginning and during the course of the trial and discussed with the investigator.
25. Requirement for continued use of CYP3A inhibitors, inducers or substrates (listed in Appendix 4).
26. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption should not take this medicine as this medicinal product contains lactose.
27. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Part A: Determine maximum tolerated dose (MTD) of palbociclib plus avelumab in advanced breast cancer | 18 month recruitment period
  Define MTD of palbociclib delivered in combination with avelumab
Part B: Determine the confirmed objective response rate of AR+ TNBC patients treated with palbociclib plus avelumab | Up to 24 month recruitment period
  Response rate assessed by RECIST 1.1 by local radiology review

SECONDARY OUTCOMES:
Determine the clinical benefit rate (CR/PR/SD for a minimum of 24 weeks) in AR+ TNBC patients treated with palbociclib plus avelumab | Total 42 month recruitment period
  Clinical benefit rate (response or stable disease lasting at least 24 weeks), assessed by RECIST 1.1 by local radiology review.
Determine the median PFS in AR+ TNBC patients treated with palbociclib plus avelumab | Total 42 month recruitment period
  Progression-free survival, calculated from day 1 of study treatment to the date of radiological disease progression or death from any cause.
Assess the safety and tolerability of palbociclib plus avelumab by recording adverse events until 30 days after the last dose of either study treatment | Total 42 month recruitment period
  Overall safety and tolerability of palbociclib with avelumab. Toxicity will be assessed by CTCAE (version 5) every 4 weeks during study treatment. Adverse events, including serious adverse events, will be recorded until 30 days after the last dose of study treatment with palbociclib or avelumab.
Assess overall survival in both parts A & B | Total 42 month recruitment period
  Overall survival, calculated from day 1 of study treatment to the date of death from any cause.

OTHER OUTCOMES:
RR in patients with PAM50 luminal archival primary tumours compared to PAM50 non luminal as a potential alternative companion diagnostic | Total 42 month recruitment period
  Objective response rate in PAM50 luminal tumours compared to PAM50 non-luminal tumours
Determine the RR in patients with PD-L1 positive compared to PDL-1 negative tumours | Total 42 month recruitment period
  Objective response rate in PDL-1 positive compared to PDL-1 negative tumours
Determine the RR in patients with high versus low mutational load | Total 42 month recruitment period
  Objective response rate in high mutational load tumours compared to low mutational load tumours
Determine the RR in patients with high tumour infiltrating lymphocytes (TILs) in the baseline and on-treatment biopsy compared to low TILs. | Total 42 month recruitment period
  Objective response rate in high TILs tumours compared to low TILs tumours at baseline and at D15
Investigate the significance of ctDNA suppression as a potential biomarker on palbociclib run-in for patients with trackable ctDNA mutations. | Total 42 month recruitment period
  Exploratory assessment of ctDNA suppression as a potential biomarker of response. Described as the proportion of patients with any suppression among the patients with the best overall response of CR or PR and the non-responders SD or PD patients the 95% CI will be reported as appropriate.
Investigate changes in peripheral blood mononuclear cells (PBMC) in patients receiving avelumab and palbociclib and the relationship with treatment response | Total 42 month recruitment period
  Exploratory assessment of tumour reactive PBMC changes between baseline, D15 and D43.
Investigate changes in T-cell and T-cell receptor clonality in patients receiving avelumab and palbociclib and the relationship with treatment response | Total 42 month recruitment period
  Exploratory assessment of dynamic changes in T-cell clonality and T-cell receptor clonality between baseline and D15 and disease progression
Evaluate potential biomarkers of sensitivity and resistance to the combination including RB1 mutations, PIK3CA mutations and loss of PTEN expression. | Total 42 month recruitment period
  Exploratory assessment of biomarkers of response in baseline tumour biopsy, and of acquired resistance in progression biopsies and plasma DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Okines, Principal Investigator — The Royal Marsden Hospital
Locations (9):
- United Kingdom (9):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Addenbrooke's Hospital Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Hope Clinical Trials Cancer Centre, Leicester
  - Barts Cancer Institute, London
  - Royal Marsden NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Nottingham University Hospital, Nottingham
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Sorlie T, Perou CM, Tibshirani R, Aas T, Geisler S, Johnsen H, Hastie T, Eisen MB, van de Rijn M, Jeffrey SS, Thorsen T, Quist H, Matese JC, Brown PO, Botstein D, Lonning PE, Borresen-Dale AL. Gene expression patterns of breast carcinomas distinguish tumor subclasses with clinical implications. Proc Natl Acad Sci U S A. 2001 Sep 11;98(19):10869-74. doi: 10.1073/pnas.191367098. PMID 11553815
- [Background] Sorlie T, Tibshirani R, Parker J, Hastie T, Marron JS, Nobel A, Deng S, Johnsen H, Pesich R, Geisler S, Demeter J, Perou CM, Lonning PE, Brown PO, Borresen-Dale AL, Botstein D. Repeated observation of breast tumor subtypes in independent gene expression data sets. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8418-23. doi: 10.1073/pnas.0932692100. Epub 2003 Jun 26. PMID 12829800
- [Background] Lehmann BD, Bauer JA, Chen X, Sanders ME, Chakravarthy AB, Shyr Y, Pietenpol JA. Identification of human triple-negative breast cancer subtypes and preclinical models for selection of targeted therapies. J Clin Invest. 2011 Jul;121(7):2750-67. doi: 10.1172/JCI45014. PMID 21633166
- [Background] Lehmann BD, Jovanovic B, Chen X, Estrada MV, Johnson KN, Shyr Y, Moses HL, Sanders ME, Pietenpol JA. Refinement of Triple-Negative Breast Cancer Molecular Subtypes: Implications for Neoadjuvant Chemotherapy Selection. PLoS One. 2016 Jun 16;11(6):e0157368. doi: 10.1371/journal.pone.0157368. eCollection 2016. PMID 27310713
- [Background] Wang C, Pan B, Zhu H, Zhou Y, Mao F, Lin Y, Xu Q, Sun Q. Prognostic value of androgen receptor in triple negative breast cancer: A meta-analysis. Oncotarget. 2016 Jul 19;7(29):46482-46491. doi: 10.18632/oncotarget.10208. PMID 27374089
- [Background] Tsang JY, Ni YB, Chan SK, Shao MM, Law BK, Tan PH, Tse GM. Androgen receptor expression shows distinctive significance in ER positive and negative breast cancers. Ann Surg Oncol. 2014 Jul;21(7):2218-28. doi: 10.1245/s10434-014-3629-2. Epub 2014 Mar 18. PMID 24639191
- [Background] McNamara KM, Yoda T, Nurani AM, Shibahara Y, Miki Y, Wang L, Nakamura Y, Suzuki K, Yang Y, Abe E, Hirakawa H, Suzuki T, Nemoto N, Miyashita M, Tamaki K, Ishida T, Brown KA, Ohuchi N, Sasano H. Androgenic pathways in the progression of triple-negative breast carcinoma: a comparison between aggressive and non-aggressive subtypes. Breast Cancer Res Treat. 2014 Jun;145(2):281-93. doi: 10.1007/s10549-014-2942-6. Epub 2014 Apr 9. PMID 24715382
- [Background] Pistelli M, Caramanti M, Biscotti T, Santinelli A, Pagliacci A, De Lisa M, Ballatore Z, Ridolfi F, Maccaroni E, Bracci R, Berardi R, Battelli N, Cascinu S. Androgen receptor expression in early triple-negative breast cancer: clinical significance and prognostic associations. Cancers (Basel). 2014 Jun 27;6(3):1351-62. doi: 10.3390/cancers6031351. PMID 24978437
- [Background] Luo X, Shi YX, Li ZM, Jiang WQ. Expression and clinical significance of androgen receptor in triple negative breast cancer. Chin J Cancer. 2010 Jun;29(6):585-90. doi: 10.5732/cjc.009.10673. PMID 20507730
- [Background] Asano Y, Kashiwagi S, Onoda N, Kurata K, Morisaki T, Noda S, Takashima T, Ohsawa M, Kitagawa S, Hirakawa K. Clinical verification of sensitivity to preoperative chemotherapy in cases of androgen receptor-expressing positive breast cancer. Br J Cancer. 2016 Jan 12;114(1):14-20. doi: 10.1038/bjc.2015.434. PMID 26757422
- [Background] Gucalp A, Tolaney S, Isakoff SJ, Ingle JN, Liu MC, Carey LA, Blackwell K, Rugo H, Nabell L, Forero A, Stearns V, Doane AS, Danso M, Moynahan ME, Momen LF, Gonzalez JM, Akhtar A, Giri DD, Patil S, Feigin KN, Hudis CA, Traina TA; Translational Breast Cancer Research Consortium (TBCRC 011). Phase II trial of bicalutamide in patients with androgen receptor-positive, estrogen receptor-negative metastatic Breast Cancer. Clin Cancer Res. 2013 Oct 1;19(19):5505-12. doi: 10.1158/1078-0432.CCR-12-3327. Epub 2013 Aug 21. PMID 23965901
- [Background] Traina TA, Miller K, Yardley DA, Eakle J, Schwartzberg LS, O'Shaughnessy J, Gradishar W, Schmid P, Winer E, Kelly C, Nanda R, Gucalp A, Awada A, Garcia-Estevez L, Trudeau ME, Steinberg J, Uppal H, Tudor IC, Peterson A, Cortes J. Enzalutamide for the Treatment of Androgen Receptor-Expressing Triple-Negative Breast Cancer. J Clin Oncol. 2018 Mar 20;36(9):884-890. doi: 10.1200/JCO.2016.71.3495. Epub 2018 Jan 26. PMID 29373071
- [Background] Bonnefoi H, Grellety T, Tredan O, Saghatchian M, Dalenc F, Mailliez A, L'Haridon T, Cottu P, Abadie-Lacourtoisie S, You B, Mousseau M, Dauba J, Del Piano F, Desmoulins I, Coussy F, Madranges N, Grenier J, Bidard FC, Proudhon C, MacGrogan G, Orsini C, Pulido M, Goncalves A. A phase II trial of abiraterone acetate plus prednisone in patients with triple-negative androgen receptor positive locally advanced or metastatic breast cancer (UCBG 12-1). Ann Oncol. 2016 May;27(5):812-8. doi: 10.1093/annonc/mdw067. Epub 2016 Feb 18. PMID 27052658
- [Background] Musgrove EA, Caldon CE, Barraclough J, Stone A, Sutherland RL. Cyclin D as a therapeutic target in cancer. Nat Rev Cancer. 2011 Jul 7;11(8):558-72. doi: 10.1038/nrc3090. PMID 21734724
- [Background] Malumbres M, Barbacid M. Cell cycle, CDKs and cancer: a changing paradigm. Nat Rev Cancer. 2009 Mar;9(3):153-66. doi: 10.1038/nrc2602. PMID 19238148
- [Background] Aarts M, Linardopoulos S, Turner NC. Tumour selective targeting of cell cycle kinases for cancer treatment. Curr Opin Pharmacol. 2013 Aug;13(4):529-35. doi: 10.1016/j.coph.2013.03.012. Epub 2013 Apr 15. PMID 23597425
- [Background] Sherr CJ, Roberts JM. CDK inhibitors: positive and negative regulators of G1-phase progression. Genes Dev. 1999 Jun 15;13(12):1501-12. doi: 10.1101/gad.13.12.1501. No abstract available. PMID 10385618
- [Background] Finn RS, Dering J, Conklin D, Kalous O, Cohen DJ, Desai AJ, Ginther C, Atefi M, Chen I, Fowst C, Los G, Slamon DJ. PD 0332991, a selective cyclin D kinase 4/6 inhibitor, preferentially inhibits proliferation of luminal estrogen receptor-positive human breast cancer cell lines in vitro. Breast Cancer Res. 2009;11(5):R77. doi: 10.1186/bcr2419. PMID 19874578
- [Background] Cancer Genome Atlas Network. Comprehensive molecular portraits of human breast tumours. Nature. 2012 Oct 4;490(7418):61-70. doi: 10.1038/nature11412. Epub 2012 Sep 23. PMID 23000897
- [Background] Asghar U, Witkiewicz AK, Turner NC, Knudsen ES. The history and future of targeting cyclin-dependent kinases in cancer therapy. Nat Rev Drug Discov. 2015 Feb;14(2):130-46. doi: 10.1038/nrd4504. PMID 25633797
- [Background] Asghar US, Barr AR, Cutts R, Beaney M, Babina I, Sampath D, Giltnane J, Lacap JA, Crocker L, Young A, Pearson A, Herrera-Abreu MT, Bakal C, Turner NC. Single-Cell Dynamics Determines Response to CDK4/6 Inhibition in Triple-Negative Breast Cancer. Clin Cancer Res. 2017 Sep 15;23(18):5561-5572. doi: 10.1158/1078-0432.CCR-17-0369. Epub 2017 Jun 12. PMID 28606920
- [Background] Goel S, DeCristo MJ, Watt AC, BrinJones H, Sceneay J, Li BB, Khan N, Ubellacker JM, Xie S, Metzger-Filho O, Hoog J, Ellis MJ, Ma CX, Ramm S, Krop IE, Winer EP, Roberts TM, Kim HJ, McAllister SS, Zhao JJ. CDK4/6 inhibition triggers anti-tumour immunity. Nature. 2017 Aug 24;548(7668):471-475. doi: 10.1038/nature23465. Epub 2017 Aug 16. PMID 28813415
- [Background] Hurvitz S MM, Fernandez Abad M, Chan D, Rostorfer R, Petru E, Barriga S, Costigan TM Michael, Caldwell CW William, Nguyen T, Press M and Slamon D, editor Biological effects of abemaciclib in a phase 2 neoadjuvant study for postmenopausal patients with HR+, HER2- breast cancer. 2016 San Antonio Breast Cancer Symposium; 2016; San Antonio, Texas
- [Background] Mittendorf EA, Philips AV, Meric-Bernstam F, Qiao N, Wu Y, Harrington S, Su X, Wang Y, Gonzalez-Angulo AM, Akcakanat A, Chawla A, Curran M, Hwu P, Sharma P, Litton JK, Molldrem JJ, Alatrash G. PD-L1 expression in triple-negative breast cancer. Cancer Immunol Res. 2014 Apr;2(4):361-70. doi: 10.1158/2326-6066.CIR-13-0127. Epub 2014 Jan 10. PMID 24764583
- [Background] Denkert C, von Minckwitz G, Darb-Esfahani S, Lederer B, Heppner BI, Weber KE, Budczies J, Huober J, Klauschen F, Furlanetto J, Schmitt WD, Blohmer JU, Karn T, Pfitzner BM, Kummel S, Engels K, Schneeweiss A, Hartmann A, Noske A, Fasching PA, Jackisch C, van Mackelenbergh M, Sinn P, Schem C, Hanusch C, Untch M, Loibl S. Tumour-infiltrating lymphocytes and prognosis in different subtypes of breast cancer: a pooled analysis of 3771 patients treated with neoadjuvant therapy. Lancet Oncol. 2018 Jan;19(1):40-50. doi: 10.1016/S1470-2045(17)30904-X. Epub 2017 Dec 7. PMID 29233559
- [Background] Kashiwagi S, Asano Y, Goto W, Takada K, Takahashi K, Noda S, Takashima T, Onoda N, Tomita S, Ohsawa M, Hirakawa K, Ohira M. Use of Tumor-infiltrating lymphocytes (TILs) to predict the treatment response to eribulin chemotherapy in breast cancer. PLoS One. 2017 Feb 6;12(2):e0170634. doi: 10.1371/journal.pone.0170634. eCollection 2017. PMID 28166544
- [Background] Nanda R, Chow LQ, Dees EC, Berger R, Gupta S, Geva R, Pusztai L, Pathiraja K, Aktan G, Cheng JD, Karantza V, Buisseret L. Pembrolizumab in Patients With Advanced Triple-Negative Breast Cancer: Phase Ib KEYNOTE-012 Study. J Clin Oncol. 2016 Jul 20;34(21):2460-7. doi: 10.1200/JCO.2015.64.8931. Epub 2016 May 2. PMID 27138582
- [Background] Fry DW, Harvey PJ, Keller PR, Elliott WL, Meade M, Trachet E, Albassam M, Zheng X, Leopold WR, Pryer NK, Toogood PL. Specific inhibition of cyclin-dependent kinase 4/6 by PD 0332991 and associated antitumor activity in human tumor xenografts. Mol Cancer Ther. 2004 Nov;3(11):1427-38. PMID 15542782
- [Background] Dean JL, McClendon AK, Hickey TE, Butler LM, Tilley WD, Witkiewicz AK, Knudsen ES. Therapeutic response to CDK4/6 inhibition in breast cancer defined by ex vivo analyses of human tumors. Cell Cycle. 2012 Jul 15;11(14):2756-61. doi: 10.4161/cc.21195. Epub 2012 Jul 15. PMID 22767154
- [Background] Finn RS, Crown JP, Lang I, Boer K, Bondarenko IM, Kulyk SO, Ettl J, Patel R, Pinter T, Schmidt M, Shparyk Y, Thummala AR, Voytko NL, Fowst C, Huang X, Kim ST, Randolph S, Slamon DJ. The cyclin-dependent kinase 4/6 inhibitor palbociclib in combination with letrozole versus letrozole alone as first-line treatment of oestrogen receptor-positive, HER2-negative, advanced breast cancer (PALOMA-1/TRIO-18): a randomised phase 2 study. Lancet Oncol. 2015 Jan;16(1):25-35. doi: 10.1016/S1470-2045(14)71159-3. Epub 2014 Dec 16. PMID 25524798
- [Background] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613
- [Background] Turner NC, Huang Bartlett C, Cristofanilli M. Palbociclib in Hormone-Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2015 Oct 22;373(17):1672-3. doi: 10.1056/NEJMc1510345. No abstract available. PMID 26488700
- [Background] Heery CR, O'Sullivan-Coyne G, Madan RA, Cordes L, Rajan A, Rauckhorst M, Lamping E, Oyelakin I, Marte JL, Lepone LM, Donahue RN, Grenga I, Cuillerot JM, Neuteboom B, Heydebreck AV, Chin K, Schlom J, Gulley JL. Avelumab for metastatic or locally advanced previously treated solid tumours (JAVELIN Solid Tumor): a phase 1a, multicohort, dose-escalation trial. Lancet Oncol. 2017 May;18(5):587-598. doi: 10.1016/S1470-2045(17)30239-5. Epub 2017 Mar 31. PMID 28373007
- [Background] Apolo AB, Infante JR, Balmanoukian A, Patel MR, Wang D, Kelly K, Mega AE, Britten CD, Ravaud A, Mita AC, Safran H, Stinchcombe TE, Srdanov M, Gelb AB, Schlichting M, Chin K, Gulley JL. Avelumab, an Anti-Programmed Death-Ligand 1 Antibody, In Patients With Refractory Metastatic Urothelial Carcinoma: Results From a Multicenter, Phase Ib Study. J Clin Oncol. 2017 Jul 1;35(19):2117-2124. doi: 10.1200/JCO.2016.71.6795. Epub 2017 Apr 4. PMID 28375787
- [Background] Patel MR, Ellerton J, Infante JR, Agrawal M, Gordon M, Aljumaily R, Britten CD, Dirix L, Lee KW, Taylor M, Schoffski P, Wang D, Ravaud A, Gelb AB, Xiong J, Rosen G, Gulley JL, Apolo AB. Avelumab in metastatic urothelial carcinoma after platinum failure (JAVELIN Solid Tumor): pooled results from two expansion cohorts of an open-label, phase 1 trial. Lancet Oncol. 2018 Jan;19(1):51-64. doi: 10.1016/S1470-2045(17)30900-2. Epub 2017 Dec 5. PMID 29217288
- [Background] Gulley JL, Rajan A, Spigel DR, Iannotti N, Chandler J, Wong DJL, Leach J, Edenfield WJ, Wang D, Grote HJ, Heydebreck AV, Chin K, Cuillerot JM, Kelly K. Avelumab for patients with previously treated metastatic or recurrent non-small-cell lung cancer (JAVELIN Solid Tumor): dose-expansion cohort of a multicentre, open-label, phase 1b trial. Lancet Oncol. 2017 May;18(5):599-610. doi: 10.1016/S1470-2045(17)30240-1. Epub 2017 Mar 31. PMID 28373005
- [Background] Dirix LY, Takacs I, Jerusalem G, Nikolinakos P, Arkenau HT, Forero-Torres A, Boccia R, Lippman ME, Somer R, Smakal M, Emens LA, Hrinczenko B, Edenfield W, Gurtler J, von Heydebreck A, Grote HJ, Chin K, Hamilton EP. Avelumab, an anti-PD-L1 antibody, in patients with locally advanced or metastatic breast cancer: a phase 1b JAVELIN Solid Tumor study. Breast Cancer Res Treat. 2018 Feb;167(3):671-686. doi: 10.1007/s10549-017-4537-5. Epub 2017 Oct 23. PMID 29063313
- [Background] Kaufman HL, Russell JS, Hamid O, Bhatia S, Terheyden P, D'Angelo SP, Shih KC, Lebbe C, Milella M, Brownell I, Lewis KD, Lorch JH, von Heydebreck A, Hennessy M, Nghiem P. Updated efficacy of avelumab in patients with previously treated metastatic Merkel cell carcinoma after >/=1 year of follow-up: JAVELIN Merkel 200, a phase 2 clinical trial. J Immunother Cancer. 2018 Jan 19;6(1):7. doi: 10.1186/s40425-017-0310-x. PMID 29347993
- [Background] Kaufman HL, Russell J, Hamid O, Bhatia S, Terheyden P, D'Angelo SP, Shih KC, Lebbe C, Linette GP, Milella M, Brownell I, Lewis KD, Lorch JH, Chin K, Mahnke L, von Heydebreck A, Cuillerot JM, Nghiem P. Avelumab in patients with chemotherapy-refractory metastatic Merkel cell carcinoma: a multicentre, single-group, open-label, phase 2 trial. Lancet Oncol. 2016 Oct;17(10):1374-1385. doi: 10.1016/S1470-2045(16)30364-3. Epub 2016 Sep 1. PMID 27592805
- [Background] Herrera-Abreu MT, Palafox M, Asghar U, Rivas MA, Cutts RJ, Garcia-Murillas I, Pearson A, Guzman M, Rodriguez O, Grueso J, Bellet M, Cortes J, Elliott R, Pancholi S, Baselga J, Dowsett M, Martin LA, Turner NC, Serra V. Early Adaptation and Acquired Resistance to CDK4/6 Inhibition in Estrogen Receptor-Positive Breast Cancer. Cancer Res. 2016 Apr 15;76(8):2301-13. doi: 10.1158/0008-5472.CAN-15-0728. Epub 2016 Mar 28. PMID 27020857
- [Background] Schaer DA, Beckmann RP, Dempsey JA, Huber L, Forest A, Amaladas N, Li Y, Wang YC, Rasmussen ER, Chin D, Capen A, Carpenito C, Staschke KA, Chung LA, Litchfield LM, Merzoug FF, Gong X, Iversen PW, Buchanan S, de Dios A, Novosiadly RD, Kalos M. The CDK4/6 Inhibitor Abemaciclib Induces a T Cell Inflamed Tumor Microenvironment and Enhances the Efficacy of PD-L1 Checkpoint Blockade. Cell Rep. 2018 Mar 13;22(11):2978-2994. doi: 10.1016/j.celrep.2018.02.053. PMID 29539425